CLINICAL TRIAL: NCT00310856
Title: A Phase 2, Partially Randomized, Open Label, Multicenter Study to Evaluate the Safety and Immunogenicity After One or Two Doses of Novartis (Formerly Chiron) Meningococcal ACWY Conjugate Vaccine Administered to Healthy Infants and Young Children
Brief Title: Immunogenicity and Safety of MenACWY in Infants (6 & 12 Months)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59P9
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Meningococcal Meningitis
Keywords: meningitis; children; vaccine
MeSH Terms: conditions — Meningitis, Meningococcal; Meningitis | interventions — MenACWY-CRM vaccine; MenC-CRM vaccine; serogroup C meningococcal conjugate vaccine; diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine; Tetanus Toxoid; pentacel; Heptavalent Pneumococcal Conjugate Vaccine

ARMS (3):
- MenACWY-CRM_6-12 M (Experimental): Subjects received 2 doses of MenACWY-CRM (1 dose at 6 and 12 months of age). Subjects also received routine vaccines: 2 doses of PC7 (1 dose at 6 and 12 months of age), 1 dose of DTaP-Hib-IPV (at 6 months of age) and 1 dose of MMR+Varicella (at 13 months of age)
  Interventions: Biological: MenACWY-CRM; Biological: DTaP-Hib-IPV; Biological: PC7; Biological: MMR; Biological: Varicella
- MenACWY-CRM_12 M (Experimental): Subjects received 1 dose of MenACWY-CRM at 12 months of age. Subjects also received routine vaccines: 2 doses of PC7 (1 dose at 6 and 12 months of age), 1 dose of DTaP-Hib-IPV (at 6 months of age) and 1 dose of MMR+Varicella (at 13 months of age)
  Interventions: Biological: MenACWY-CRM; Biological: DTaP-Hib-IPV; Biological: PC7; Biological: MMR; Biological: Varicella
- MenC-CRM_12 M_MenACWY-CRM_18 M (Experimental): Subjects received 1 dose of MenC-CRM (at 12 months of age) and 1 dose of MenACWY-CRM (at 18 months of age).
  Subjects also received routine vaccines: 1 dose of PCV7 (at 12 months), MMR+Varicella (at 13 months) and DTaP-Hib-IPV (at 18 months)
  Interventions: Biological: MenACWY-CRM; Biological: MenC-CRM; Biological: DTaP-Hib-IPV; Biological: PC7; Biological: MMR; Biological: Varicella

INTERVENTIONS:
Biological: MenACWY-CRM — Subjects received the full dose (0.5 mL) of MenACWY-CRM, obtained by extemporaneous mixing of lyophilized MenA powder component and the MenCWY suspension, administered by IM injection into the anterolateral area of the right thigh.
  Other Names: Meningococcal ACWY conjugate vaccine
Biological: MenC-CRM — One dose (0.5 mL) of MenC-CRM was obtained by extemporaneous mixing just before injection of the lyophilized MenC component and a saline solvent, administered by IM injection into the arm region.
  Other Names: Meningococcal C conjugate vaccine
  Arms: MenC-CRM_12 M_MenACWY-CRM_18 M
Biological: DTaP-Hib-IPV
  Other Names: Combined vaccine containing diphtheria, tetanus, pertussis, Haemophilus influenzae type B and inactivated polio virus; Pentacel
Biological: PC7 — One dose (0.5 mL) of PC7, supplied in pre-filled syringe, administered by IM injection into the anterolateral area of the left thigh.
  Other Names: Heptavalent conjugate pneumococcal; Prevnar
Biological: MMR
  Other Names: Measles, mumps and rubella
Biological: Varicella

SUMMARY:
To assess the immunogenicity of Novartis (formerly Chiron) Meningococcal ACWY conjugate vaccine (MenACWY) when administered as a two-dose schedule at 6 and 12 months of age.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for Groups I (MenACWY-CRM_6-12 M) and II (MenACWY-CRM_12 M)

Subjects eligible for enrollment in the study were healthy infants:

1. who were 6 months old and who were born after full-term pregnancy with an estimated gestational age of 37 weeks or greater and a birth weight 2.5 kg or greater;
2. who previously received two doses of PC7 and DTaP-Hib-IPV vaccines;
3. for whom a parent/legal guardian gave written informed consent, after the nature of the study was explained;
4. who were available for all the visits scheduled in the study;
5. who were in good health as determined by medical history, physical examination, and clinical judgment of the investigator.

Inclusion criteria for Group III (MenC-CRM_12 M_MenACWY-CRM_18 M)

Subjects eligible for enrollment in the study were healthy infants:

1. who were 12 months old;
2. who previously received three doses of DTaP-Hib-IPV (Pentacel) vaccines;
3. for whom a parent/legal guardian gave written informed consent, after the nature of the study was explained;
4. who were available for all the visits scheduled in the study;
5. who were in good health as determined by medical history, physical examination, and clinical judgment of the investigator.

Exclusion criteria:

Subjects were not to be included in this study if:

1. their parents/legal guardians were unwilling or unable to give written informed consent to participate in the study;
2. they previously received any meningococcal vaccine;
3. they had a previously ascertained or suspected disease caused by Neisseria meningitidis (N meningitidis);
4. they had a history of any anaphylactic shock, asthma, urticaria, or other allergic reaction after previous vaccinations or known hypersensitivity to any vaccine component;
5. they had experienced significant acute or chronic infection within the previous 7 days or had experienced fever (38.0ºC or greater) within the previous 3 days;
6. they had any present or suspected serious acute disease (e.g., leukemia, lymphomas), or chronic disease (e.g., with signs of cardiac failure, renal failure, severe malnutrition, or insulin-dependent diabetes), or progressive neurological disease, or a genetic anomaly/known cytogenic disorders (e.g., Down's syndrome), or who had a diagnosed cardiac defect or abnormality of hemodynamic significance (e.g., ventricular septal defect, patent ductus arteriosus, or atrial septal defect);
7. they had a known or suspected autoimmune disease or impairment /alteration of immune function resulting from use of (for example):

   * any immunosuppressive therapy since birth;
   * immunostimulants since birth;
   * any systemic corticosteroid administered for more than 5 days or in a daily dose of greater than 1 mg/kg/day prednisone or equivalent for 5 days or less in the previous 30 days;
8. they had a suspected or known HIV infection or HIV-related disease;
9. they had received parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within the past 90 days and were expected to receive it for the full length of the study;
10. they had a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time;
11. they had a history of seizure disorder:

    * febrile seizure;
    * any other seizure disorder;
12. they had taken systemic antibiotics (either oral or parenteral) within the previous 14 days (EXCEPTION: subjects who had received an oral or parenteral β-lactam antibiotic [e.g.: penicillin, amoxicillin, ceftriaxone, cefuroxime or cephalexin] could have been enrolled 7 days following the last dose);
13. their parents/legal guardians were planning to leave the area of the study center before the end of the study period;
14. they had any condition which, in the opinion of the investigator, might have interfered with the evaluation of the study objectives.

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2005-06; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Halperin, Dr., Principal Investigator — Novartis Vaccines & Diagnostics; Francisco Diaz-Mitoma, Dr., Principal Investigator — Novartis Vaccines
Locations (3):
- Canada (3):
  - Children's Hospital of Eastern Ontario Research Institute, Ottawa, Ontario
  - Herridge Community Health Clinic, Ottawa, Ontario
  - Clinical Trials Research Center, Department of Pediatrics, Dalhousie University, IWK Health Center, Halifax

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at three sites in Canada.
Pre-assignment Details: All enrolled subjects were included in the study.
Period: Overall Study
Arm/Group | MenACWY-CRM_6-12 M | MenACWY-CRM_12 M | MenC-CRM_12 M_MenACWY-CRM_18 M
Started | 64 | 61 | 50
Completed | 59 | 56 | 42
Not Completed | 5 | 5 | 8
Not completed — Withdrawal by Subject | 2 | 2 | 2
Not completed — Lost to Follow-up | 1 | 2 | 6
Not completed — Inappropriate enrollment | 1 | 1 | 0
Not completed — Unable to classify | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was done for all enrolled subjects.
Groups:
- MenACWY-CRM_6-12 M: Subjects received 2 doses of MenACWY-CRM at 6 and 12 months of age. Subjects also received routine vaccines: 2 doses of PC7 (at 6 and 12 months) and 1 dose each of DTaP-Hib-IPV (at 6 months) and MMR+Varicella (at 13 months).
- MenACWY-CRM_12 M: Subjects received 1 dose of MenACWY-CRM at 12 months of age. Subjects also received routine vaccines: 2 doses of PC7 (at 6 and 12 months) and 1 dose each of DTaP-Hib-IPV (at 6 months) and MMR+Varicella (at 13 months).
- MenC-CRM_12 M_MenACWY-CRM_18 M: Subjects received 1 dose each of MenC-CRM (at 12 months) and MenACWY-CRM (at 12 months).
  Subjects also received routine vaccines: 1 dose each of PC7 (at 12 months), MMR+Varicella (at 13 months) and DTaP-Hib-IPV (at 18 months).
- Total: Total of all reporting groups
Arm/Group | MenACWY-CRM_6-12 M | MenACWY-CRM_12 M | MenC-CRM_12 M_MenACWY-CRM_18 M | Total
Number analyzed (Participants) | 64 | 61 | 50 | 175
Age, Continuous [Mean (Standard Deviation); unit: Months] | 6.0 (0.2) | 6.0 (0.0) | 12.1 (0.2) | 7.7 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 31 | 21 | 77
  Male | 39 | 30 | 29 | 98

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With hSBA Titers ≥1:4 Against Each of 4 Meningococcal Serogroups After MenACWY-CRM Vaccination Administered as 2-Dose or 1-Dose Schedule
Description: Immunogenicity was measured as the percentage of subjects with hSBA titers ≥1:4 against meningococcal serogroups A, C, W and Y, evaluated by serum bactericidal assay using human complement (hSBA), before vaccination and 1 month after 2-dose schedule of MenACWY-CRM administered at 6 and 12 months of age (MenACWY-CRM_6-12 M group) or 1-dose schedule administered at 12 months (MenACWY-CRM_12 M group)
Time Frame: Before and 1 month after 2-dose or 1-dose schedule
Population: Analysis was done on per protocol (PP) population, i.e subjects in the exposed population who received all the relevant doses of vaccines correctly; and provided evaluable serum samples at the relevant time points; and had no major protocol violation as defined prior to unblinding.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY-CRM_6-12 M | MenACWY-CRM_12 M
Number analyzed (Participants) | 55 | 54
Percentage of subjects
  Serogroup A - Prevaccination (N=50,53) | 10 [3 to 22] | 0 [0 to 7]
  Serogroup A - Postvaccination (N=50,53) | 88 [76 to 95] | 74 [60 to 85]
  Serogroup C - Prevaccination | 85 [73 to 94] | 2 [0.047 to 10]
  Serogroup C - Postvaccination | 100 [94 to 100] | 96 [87 to 100]
  Serogroup W - Prevaccination (N=40,41) | 85 [70 to 94] | 2 [0.062 to 13]
  Serogroup W - Postvaccination (N=40,41) | 100 [91 to 100] | 95 [83 to 99]
  Serogroup Y - Prevaccination (N=53,54) | 72 [58 to 83] | 0 [0 to 7]
  Serogroup Y - Postvaccination (N=53,54) | 100 [93 to 100] | 78 [64 to 88]

2. Secondary Outcome: Geometric Mean hSBA Titers Against Each of 4 Meningococcal Serogroups After MenACWY-CRM Vaccination Administered as 2-Dose or 1-Dose Schedule
Description: The immune response was measured as the hSBA geometric mean titers (GMTs) against meningococcal serogroups A, C, W and Y, before vaccination and 1 month after 2-dose schedule of MenACWY-CRM administered at 6 and 12 months of age (MenACWY-CRM_6-12 M group) or 1-dose schedule administered at 12 months of age (MenACWY-CRM_12 M group)
Time Frame: Before and 1 month after 2-dose or 1-dose schedule
Population: Analysis was done on PP population.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titers
Arm/Group | MenACWY-CRM_6-12 M | MenACWY-CRM_12 M
Number analyzed (Participants) | 55 | 54
Geometric mean titers
  Serogroup A - Prevaccination (N=50,53) | 2.41 [2.18 to 2.65] | 1.99 [1.81 to 2.19]
  Serogroup A - Postvaccination (N=50,53) | 44 [29 to 65] | 11 [7.55 to 16]
  Serogroup C - Prevaccination | 19 [14 to 25] | 2.06 [1.54 to 2.77]
  Serogroup C - Postvaccination | 302 [224 to 405] | 40 [30 to 54]
  Serogroup W - Prevaccination (N=40,41) | 15 [12 to 19] | 2.09 [1.68 to 2.6]
  Serogroup W-Postvaccination (N=40,41) | 220 [155 to 313] | 30 [21 to 43]
  Serogroup Y - Prevaccination | 7.91 [6.64 to 9.43] | 2.02 [1.7 to 2.4]
  Serogroup Y - Postvaccination | 136 [100 to 185] | 10 [7.68 to 14]

3. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥1:8 Against Each of 4 Meningococcal Serogroups After MenACWY-CRM Vaccination Administered as 2-Dose or 1-Dose Schedule
Description: Immunogenicity was measured as the percentage of subjects with hSBA titers ≥1:8 against meningococcal serogroups A, C, W and Y, before vaccination and 1 month after 2-dose schedule of MenACWY-CRM administered at 6 and 12 months of age (MenACWY-CRM_6-12 M group) or 1-dose schedule administered at 12 months of age (MenACWY-CRM_12 M)
Time Frame: Before and 1 month after 2-dose or 1-dose schedule
Population: Analysis was done on PP population.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY-CRM_6-12 M | MenACWY-CRM_12 M
Number analyzed (Participants) | 55 | 54
Percentage of subjects
  Serogroup A - Prevaccination (N=50,53) | 8 [2 to 19] | 0 [0 to 7]
  Serogroup A - Postvaccination (N=50,53) | 84 [71 to 93] | 60 [46 to 74]
  Serogroup C - Prevaccination | 75 [61 to 85] | 2 [0.047 to 10]
  Serogroup C - Postvaccination | 100 [94 to 100] | 93 [82 to 98]
  Serogroup W - Prevaccination (N=40,41) | 73 [56 to 85] | 2 [0.062 to 13]
  Serogroup W - Postvaccination (N=40,41) | 100 [91 to 100] | 93 [80 to 98]
  Serogroup Y - Prevaccination (N=53,54) | 55 [40 to 68] | 0 [0 to 7]
  Serogroup Y - Postvaccination (N=53,54) | 100 [93 to 100] | 67 [53 to 79]

4. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥1:4 or ≥1:8 Against Meningococcal Serogroup C After One Vaccination of MenC-CRM Administered at 12 Months of Age
Description: Immunogenicity was measured as the percentage of subjects who achieved hSBA titers ≥1:4 or ≥1:8 against meningococcal serogroup C, before and 1 month after one vaccination of MenC-CRM administered concomitantly with Prevnar at 12 months of age
Time Frame: Before and 1 month after MenC-CRM vaccination at 12 months
Population: Analysis was done on PP population.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenC-CRM_12 M_MenACWY-CRM_18 M
Number analyzed (Participants) | 40
Percentage of subjects
  hSBA titers ≥1:4 - Prevaccination | 0 [0 to 9]
  hSBA titers ≥1:4 - Postvaccination | 93 [80 to 98]
  hSBA titers ≥1:8 - Prevaccination | 0 [0 to 9]
  hSBA titers ≥1:8 - Postvaccination | 88 [73 to 96]

5. Secondary Outcome: Geometric Mean hSBA Titers Against Meningococcal Serogroup C After One Vaccination of MenC-CRM Administered at 12 Months of Age
Description: The immune response was measured as the hSBA GMT against meningococcal serogroup C, before and 1 month after one vaccination of MenC-CRM administered concomitantly with Prevnar at 12 months of age
Time Frame: Before and 1 month after MenC-CRM vaccination at 12 months
Population: Analysis was done on PP population.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titers
Arm/Group | MenC-CRM_12 M_MenACWY-CRM_18 M
Number analyzed (Participants) | 40
Geometric mean titers
  hSBA GMTs - Prevaccination | 2 [1.81 to 2.21]
  hSBA GMTs - Postvaccination | 39 [29 to 52]

6. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥1:4 or ≥1:8 Against Meningococcal Serogroup A, W and Y After One Vaccination of MenACWY-CRM Administered at 18 Months of Age
Description: Immunogenicity was measured as the percentage of subjects who achieved hSBA titers ≥1:4 or ≥1:8 against meningococcal serogroups A, W and Y, before and 1 month after one vaccination of MenACWY-CRM administered concomitantly with Pentacel at 18 months of age
Time Frame: Before and 1 month after MenACWY-CRM vaccination at 18 months
Population: Analysis was done on PP population.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenC-CRM_12 M_MenACWY-CRM_18 M
Number analyzed (Participants) | 38
Percentage of subjects
  Serogroup A - hSBA ≥1:4 - Prevaccination | 0 [0 to 9]
  Serogroup A - hSBA ≥1:4 - Postvaccination | 63 [46 to 78]
  Serogroup W - hSBA ≥1:4 - Prevaccination (N=37) | 3 [0.068 to 14]
  Serogroup W - hSBA ≥1:4 - Postvaccination (N=37) | 81 [65 to 92]
  Serogroup Y - hSBA ≥1:4 - Prevaccination | 0 [0 to 9]
  Serogroup Y - hSBA ≥1:4 - Postvaccination | 79 [63 to 90]
  Serogroup A - hSBA ≥1:8 - Prevaccination | 0 [0 to 9]
  Serogroup A - hSBA ≥1:8 - Postvaccination | 50 [33 to 67]
  Serogroup W - hSBA ≥1:8 - Prevaccination (N=37) | 3 [0.068 to 14]
  Serogroup W - hSBA ≥1:8 - Postvaccination (N=37) | 76 [59 to 88]
  Serogroup Y - hSBA ≥1:8 - Prevaccination | 0 [0 to 9]
  Serogroup Y - hSBA ≥1:8 - Postvaccination | 63 [46 to 78]

7. Secondary Outcome: hSBA GMTs Against Meningococcal Serogroups A, W and Y After One Vaccination of MenACWY-CRM Administered at 18 Months of Age
Description: The immune response was measured as the hSBA GMTs against meningococcal serogroups A, W and Y, before and 1 month after one vaccination of MenACWY-CRM administered concomitantly with Pentacel at 18 months of age
Time Frame: Before and 1 month after MenACWY-CRM vaccination at 18 months
Population: Analysis was done on PP population.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titers
Arm/Group | MenC-CRM_12 M_MenACWY-CRM_18 M
Number analyzed (Participants) | 38
Geometric mean titers
  Serogroup A - Prevaccination | 2 [1.78 to 2.24]
  Serogroup A - Postvaccination | 8.05 [5.11 to 13]
  Serogroup W - Prevaccination (N=37) | 2.09 [1.66 to 2.64]
  Serogroup W - Postvaccination (N=37) | 17 [12 to 24]
  Serogroup Y - Prevaccination | 2 [1.62 to 2.45]
  Serogroup Y - Postvaccination | 13 [8.78 to 18]

8. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥1:4 or ≥1:8 Against Meningococcal Serogroup C After MenACWY-CRM Vaccination Administered at 18 Months of Age, Following One Vaccination of MenC-CRM at 12 Months of Age
Description: Booster response was measured as the percentage of subjects who achieved hSBA titers ≥1:4 or ≥1:8 against meningococcal serogroup C, before and 1 month after MenACWY-CRM vaccination administered at 18 months of age, following one vaccination of MenC-CRM at 12 months of age
Time Frame: Before and 1 month after MenACWY-CRM vaccination at 18 months
Population: Analysis was done on PP population.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenC-CRM_12 M_MenACWY-CRM_18 M
Number analyzed (Participants) | 38
Percentage of subjects
  hSBA ≥1:4 - Prevaccination | 89 [75 to 97]
  hSBA ≥1:4 - Postvaccination | 100 [91 to 100]
  hSBA ≥1:8 - Prevaccination | 82 [66 to 92]
  hSBA ≥1:8 - Postvaccination | 100 [91 to 100]

9. Secondary Outcome: hSBA GMT Against Meningococcal Serogroup C After MenACWY-CRM Vaccination Administered at 18 Months of Age, Following One Vaccination of MenC-CRM at 12 Months of Age
Description: Booster response was measured as the hSBA GMT against meningococcal serogroup C, before and 1 month after MenACWY-CRM vaccination administered at 18 months of age, following one vaccination of MenC-CRM at 12 months of age
Time Frame: Before and 1 month after MenACWY-CRM vaccination at 18 months
Population: Analysis was done on PP population.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titers
Arm/Group | MenC-CRM_12 M_MenACWY-CRM_18 M
Number analyzed (Participants) | 38
Geometric mean titers
  hSBA GMTs - Prevaccination | 29 [20 to 41]
  hSBA GMTs - Postvaccination | 667 [467 to 952]

10. Secondary Outcome: Number of Subjects Who Reported Solicited Local and Systemic Reactions After Any MenACWY-CRM, MenC-CRM and Concomitant Vaccination
Description: The safety was assessed as the number of subjects who reported solicited local and systemic reactions from day 1 through day 7 following any vaccination of MenACWY-CRM, MenC-CRM and concomitant vaccination
Time Frame: From day 1 through day 7 after any vaccination
Population: Analysis was done on the safety population, i.e. all subjects who had at least one vaccination and some postbaseline safety data.
Measure: Number; unit: participants
Arm/Group | MenACWY-CRM_6-12 M | MenACWY-CRM_12 M | MenC-CRM_12 M_MenACWY-CRM_18 M
Number analyzed (Participants) | 64 | 61 | 50
participants
  Any local reactions | 53 | 49 | 47
  MenACWY MenC Tenderness (N=64,56,50) | 25 | 24 | 30
  MenACWY MenC Erythema (N=64,56,50) | 33 | 25 | 28
  MenACWY MenC Induration (N=64,56,50) | 29 | 20 | 23
  DTaP-Hib-IPV Tenderness (N=64,61,44) | 23 | 22 | 27
  DTaP-Hib-IPV Erythema (N=64,61,44) | 33 | 25 | 23
  DTaP-Hib-IPV Induration (N=64,61,44) | 28 | 20 | 17
  PCV7 Tenderness | 32 | 33 | 16
  PC7 Erythema | 39 | 31 | 28
  PC7 Induration | 31 | 32 | 19
  Any systemic reactions | 59 | 55 | 43
  Change in eating habits (N=62,60,50) | 28 | 21 | 21
  Sleepiness | 35 | 32 | 22
  Irritability | 57 | 45 | 38
  Vomiting | 9 | 11 | 6
  Diarrhea | 12 | 18 | 11
  Fever (≥38 °C) | 6 | 12 | 12
  Analgesic Antipyretic Medicines Used | 42 | 35 | 29

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were reported throughout the study (day 1 through day 336)
Groups:
- MenACWY-CRM_6-12M: Subjects received 2 doses of MenACWY-CRM at 6 and 12 months of age. Subjects also received routine vaccines: 2 doses of PC7 (at 6 and 12 months) and 1 dose each of DTaP-Hib-IPV (at 6 months) and MMR+Varicella (at 13 months)
- MenACWY-CRM_12M: Subjects received 1 dose of MenACWY-CRM at 12 months of age. Subjects also received routine vaccines: 2 doses of PC7 (at 6 and 12 months) and 1 dose each of DTaP-Hib-IPV (at 6 months) and MMR+Varicella (at 13 months)
- MenC-CRM_12M_MenACWY-CRM_18M: Subjects received 1 dose each of MenC-CRM (at 12 months) and MenACWY-CRM (at 12 months). Subjects also received routine vaccines: 1 dose each of PC7 (at 12 months), MMR+Varicella (at 13 months) and DTaP-Hib- IPV (at 18 months)
Arm/Group | MenACWY-CRM_6-12M | MenACWY-CRM_12M | MenC-CRM_12M_MenACWY-CRM_18M
Serious Adverse Events (participants affected / at risk) | 3/64 | 2/61 | 2/50
Other Adverse Events (participants affected / at risk) | 62/64 | 58/61 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM_6-12M (N=64) | MenACWY-CRM_12M (N=61) | MenC-CRM_12M_MenACWY-CRM_18M (N=50)
Bronchiolitis (Infections and infestations) | 1 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM_6-12M (N=64) | MenACWY-CRM_12M (N=61) | MenC-CRM_12M_MenACWY-CRM_18M (N=50)
Diarrhoea (Gastrointestinal disorders) | 12 | 18 | 13
Vomiting (Gastrointestinal disorders) | 9 | 11 | 7
Injection site erythema (General disorders) | 41 | 33 | 39
Injection site induration (General disorders) | 38 | 35 | 31
Injection site pain (General disorders) | 36 | 35 | 34
Irritability (General disorders) | 57 | 45 | 38
Pyrexia (General disorders) | 6 | 14 | 13
Nasopharyngitis (Infections and infestations) | 6 | 5 | 4
Somnolence (Nervous system disorders) | 35 | 32 | 22
Eating disorder (Psychiatric disorders) | 28 | 21 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigators from publishing. Any publications from a single site are postponed until the publication of the pool data (i.e., data from all sites) in the clinical trial.